CLINICAL TRIAL: NCT07276997
Title: A Phase 2, Multicenter, 6-Week, Double Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Icalcaprant in Subjects With Major Depressive Disorder
Brief Title: A Study to Assess Change in Disease Activity and Adverse Events of Oral Icalcaprant in Adult Participants With Major Depressive Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M25-987
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Icalcaprant
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Icalcaprant Dose A (Experimental): Participants will receive oral Icalcaprant dose A once daily for 6 weeks and attend a follow up visit 30 days following end of treatment.
  Interventions: Drug: Icalcaprant
- Icalcaprant Dose B (Experimental): Participants will receive oral Icalcaprant dose B once daily for 6 weeks and attend a follow up visit 30 days following end of treatment.
  Interventions: Drug: Icalcaprant
- Placebo for Icalcaprant (Placebo Comparator): Participants will receive oral placebo once daily for 6 weeks and attend a follow up visit 30 days following end of treatment.
  Interventions: Drug: Placebo for Icalcaprant

INTERVENTIONS:
Drug: Icalcaprant — Oral Capsules
  Arms: Icalcaprant Dose A; Icalcaprant Dose B
Drug: Placebo for Icalcaprant — Oral Capsules
  Arms: Placebo for Icalcaprant

SUMMARY:
Major depressive disorder (MDD; depression) is a mood disorder that causes a continued feeling of sadness and loss of interest. It is a common and serious illness that can cause both emotional and physical symptoms such as feelings of sadness, irritability, not being able to focus on activities, tiredness, changes in eating habits, and aches and pains. This study will assess the changes in disease activity and adverse events of oral Icalcaprant in adult participants with major depressive disorder who are currently experiencing a major depressive episode (MDE).

Icalcaprant is an investigational drug being developed for the treatment of depressive episodes in adult participants with major depressive disorder. Participants are placed in 1 of 3 groups, called treatment arms. There is a 1 in 3 chance that a participant will be assigned to placebo treatment. Around 195 adult participant with major depressive disorder will be enrolled in approximately 35 sites in North America.

Participants will receive oral capsules of Icalcaprant or matching placebo once daily for 6 weeks, with a 30-day safety follow-up.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of major depressive disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, fifth edition, text revision (DSM-5-TR) without psychotic features, confirmed by the Mini International Neuropsychiatric Interview (MINI) 7.0.
* Body Mass Index (BMI) is ≥ 18.0 to ≤ 35.0 kg/m^2
* Currently experiencing an major depressive episode (MDE) beginning at least 4 weeks prior to consent and not exceeding 6 months prior to Screening
* Normal physical examination findings, clinical laboratory test results, vital signs, and 12-lead ECG results at Visit 1 or abnormal results that are judged not clinically significant by the investigator and documented as such in the eCRF.

Exclusion Criteria:

* Has failed (no more than 25% response on Antidepressant Treatment History Questionnaire (ATRQ)) 3 or more antidepressant treatments during the current depressive episode despite an adequate dose (per ATRQ) and duration (at least 6 weeks).
* History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) total score. | Up to approximately 6 weeks
  Montgomery-Åsberg Depression Rating Scale (MADRS) The MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants are to be rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item will be scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity.
Number of Participants with Adverse Events (AEs) | Up to approximately 10 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impression (CGIS) | Up to approximately 6 weeks
  Change from Baseline in Clinical Global Impression (CGIS)-The CGIS is a single-item clinician-reported measure of severity of depression. Clinicians are asked to consider their total clinical experience with Participants with major depressive disorder (MDD) and assess how severely ill the participant has been during the past 7 days. Response options range from 1 to 7: 1 = normal to 7 = very severely ill.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (23):
- United States (23):
  - Harmonex /ID# 277517, Dothan, Alabama
  - Ima Clinical Research Phoenix (Alea) /ID# 277516, Phoenix, Arizona
  - Preferred Research Partner, Inc /ID# 279206, Little Rock, Arkansas
  - Woodland International Research Group /ID# 277605, Little Rock, Arkansas
  - Advanced Research Center /ID# 277537, Anaheim, California
  - Sun Valley Research Center /ID# 277513, Imperial, California
  - Synergy San Diego /ID# 277553, Lemon Grove, California
  - CenExel CNR /ID# 277533, Sherman Oaks, California
  - Inland Psychiatric Medical Group Inc. /ID# 279275, Temecula, California
  - Sunwise Clinical Research /ID# 277555, Walnut Creek, California
  - CenExcel Clinical Research - Main Facility /ID# 278200, Hollywood, Florida
  - Cns Healthcare - Jacksonville /ID# 277658, Jacksonville, Florida
  - GMI Florida - Central Miami Medical Institute /ID# 278218, Miami, Florida
  - Clinical Neuroscience Solutions - Orlando - East South Street /ID# 277558, Orlando, Florida
  - Trialmed /ID# 277601, Atlanta, Georgia
  - Flourish Research - Great Lakes Clinical Trials /ID# 278201, Chicago, Illinois
  - Amr Conventions Research /ID# 277547, Warrenville, Illinois
  - Redbird Research /ID# 277485, Las Vegas, Nevada
  - Manhattan Behavioral Medicine /ID# 277910, New York, New York
  - Sooner Clinical Research /ID# 277659, Oklahoma City, Oklahoma
  - CNS Healthcare - Memphis /ID# 278192, Memphis, Tennessee
  - Community Clinical Research - Austin - Cross Park Drive /ID# 277935, Austin, Texas
  - Northwest Clinical Research Center /ID# 277484, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-987